CLINICAL TRIAL: NCT03541915
Title: The Effect of Intravenous Magnesium Sulfate on Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Gynecologic Surgery
Brief Title: Magnesium Sulfate; Postoperative Nausea and Vomiting; Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Department of Anesthesiology and Pain Medicine, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2018-0066
Record Dates: First submitted 2018-05-08; First posted 2018-05-31 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Magnesium Sulfate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mg group (Experimental): 20mg/kg of magnesium sulfate will be infused after induction of anesthesia. And magnesium sulfated will be continuously infused at a rate of 15mg/kg/h during the operation.
  Interventions: Drug: Mg (magnesium sulfate)
- Control group (Placebo Comparator): Same volume of normal saline will be infused after induction of anesthesia. And the same volume of normal saline will be continuously infused at a same rate of magnesium during the operation.
  Interventions: Drug: Control (saline)

INTERVENTIONS:
Drug: Mg (magnesium sulfate) — 20mg/kg of magnesium sulfate will be infused after induction of anesthesia. And magnesium sulfated will be continuously infused at a rate of 15mg/kg/h during the operation.
  Other Names: Masi
  Arms: Mg group
Drug: Control (saline) — The same volume of normal saline will be infused after induction of anesthesia and continuously infused at the same rate of magnesium.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
Postoperative nausea and vomiting (PONV) is commonly accompanied in patients undergoing surgery under general anesthesia. The patients undergoing laparoscopic gynecologic surgery have multiple risk factors for developing PONV such as female gender, nonsmoker, postoperative opioids, and laparoscopic surgery. Thus, it is important to prevent PONV in these patients.

DETAILED DESCRIPTION:
Magnesium is a N-methyl-D-aspartate (NMDA) antagonist that is known to be effective in reducing opioid consumption and controlling postoperative pain. This opioid reducing effect can be associated with reduction of the incidence of PONV. However, the effect of magnesium on preventing PONV have not been investigated before. Thus, the investigators hypothesized that intraoperative infusion of magnesium will be effective in preventing PONV in patients undergoing laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic disease
* Female patients undergoing laparoscopic gynecologic surgery and receiving postoperative fentanyl based intravenous patient controlled analgesia (PCA), aged 20-65 years.

Exclusion Criteria:

* impaired renal or hepatic function (Glutamic Oxalacetate Transaminase [GOT]/Glutamic Pyruvate Transaminase [GPT]>50, estimated glomerular filtration rate [eGFR]<60)
* atrioventricular block, myopathies, diabetes, treated with calcium channel blockers
* History of receiving antiemetics within 1 day before surgery
* History of receiving opioids or non-steroidal anti-inflammatory drugs within 1 week of surgery
* drugs or alcohol abuse
* patients treated with isoniazid, chlorpromazine, or digoxin
* patients who cannot communicated with others or with cognitive dysfunction
* patients who cannot read informed consent

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PONV | up to postoperative 2 days
  The incidence of PONV will be measured up to postoperative 2 days.